CLINICAL TRIAL: NCT04827212
Title: An Integrated Two-Way Communication and Near-Real-Time Sensing System to Detect and Modify Daily Inactivity Among Adults Over Age 60
Brief Title: Companion: Sensor-based Two-way Communication for Physical Activity in Older Adults
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northeastern University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Dinesh John, Associate Professor, Northeastern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20-01-15; P30AG048785 (NIH)
Record Dates: First submitted 2021-03-23; First posted 2021-04-01 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Exercise; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Control group will engage in a 16-week supervised exercise program and then be followed-up after 24 weeks
- Treatment (Experimental): Treatment group will engage in a 16-week supervised exercise program and then be followed-up after 24 weeks. In addition, the Companion will be deployed in the treatment group only.
  Interventions: Behavioral: Companion

INTERVENTIONS:
Behavioral: Companion — Companion integrates wearable sensing with the smartphone to develop a behavior-aware, virtual system that uses a "human-in-the-loop" approach to enable meaningful two-way communication. Companion builds rich models of typical behavior using sensors and context sensitive ecological momentary assessment to deliver intervention components and behavior change strategies using socially engaging, contextually salient, and tailored text-message conversations in near-real-time.
  Arms: Treatment

SUMMARY:
This pilot study is a small sample (N=46) 16-week clinical trial with a follow-up after 24-weeks among sedentary adults >60 y with a BMI >25 kg/m2 to tests the impact of a hybrid artificial intelligence behavior change system (Companion) on physical activity. Participants will be randomized to a control and intervention group. All participants will engage in a proven supervised exercise program from week 1 to 16. Only the intervention group will receive Companion from week 1 to 16.

DETAILED DESCRIPTION:
This is a single site randomized clinical trial to test if if Companion improves and sustains free-living physical activity and sedentary behaviors in adults >60 y and improves health outcomes. Forty-six sedentary adults >60 y with a BMI >25 kg/m2 will be randomized to a control and intervention group. Both groups will undergo a 16-week supervised training program involving supervised training sessions 45-60 min, twice a week. The intervention group will additionally receive the two-way communication-based Companion meta intervention. Two-way communication during weeks 1 to 4, will focus on gathering information on the adult's motivations, preferences, habits, contexts, and usual behavior patterns to build typical individual behavior models. The model will be used to develop an adaptive physical active and sedentary behavior intervention prescription. Primary outcomes from Aim 1 and exploratory outcomes from Aim 2 will be measured at baseline and then after 16 and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years and above- This intervention study focusses on this population demographic.
* Participants have a body mass index greater than 25 kg/m2- This threshold for BMI is used to classify an adult as overweight or obese
* No conditions preventing participation in physical activity lasting 10 to 30 min- Such conditions will limit prescription of physical activity/exercise components of the training program and that promoted using Companion.
* Have a smart phone- The absence of a smart phone will limit the ability of remote communication with the study participant using Companion.

Exclusion Criteria:

* Engage in structured physical activity for more than 2 days/week lasting 30 min/session- Physically active participants will not be representative of typical adults >60 y. Being active prior to study participation may mask the effects of the intervention.
* Regularly use any assistive device for walking- Use of an assistive device would limit the ability to engage in prescribed physical activity. Future work can be tailored for sub-groups in the demographic being studied.
* Likely to alter medications pertaining to cardiovascular or metabolic health- Altering medications during the study will influence change in selected outcome measures.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dinesh John, PhD, Principal Investigator — Northeastern University
Locations (1):
- Northeastern Univeristy, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 participants were excluded from the study before assignment to groups. 3 chose to not continue participation and 2 were recommended to no continue participation by their personal physician. 46 participants were randomized to th control and treatment groups
Period: Baseline to 16 Weeks
Arm/Group | Control | Treatment
Started | 23 | 23
Completed | 21 | 21
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2
Period: 16 to 24 Weeks
Arm/Group | Control | Treatment
Started | 21 | 21
Completed | 18 | 17
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Treatment | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.7 (6.1) | 68.9 (6.5) | 71 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 18 | 31
  Male | 10 | 5 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 22 | 19 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 17 | 19 | 36
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/^2] | 30.5 (3.8) | 30.4 (4.9) | 30.4 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Physical Activity Hours Per Day Measured Using a Body-worn Accelerometer at Baseline
Description: Total time spent being active will be measured using a body worn motion sensor (accelerometer) during waking hours over a period of one week. Measures for each day (hours) will be averaged to obtain a representative estimate of daily habitual behavior.
Time Frame: Baseline
Population: Accelerometer data were missing for 1 participant in the control group.This results in a discrepancy with overall participant flow table which represents the number of participants with any available data.
Measure: Mean (Standard Deviation); unit: h/day
Arm/Group | Control | Treatment
Number analyzed (Participants) | 22 | 23
h/day | 1.3 (0.5) | 1.6 (0.5)
Statistical Analysis 1: Comparison: Control vs Treatment; Test type: Superiority; p = 0.037, Mixed Models Analysis — P<0.05; Mean Difference (Final Values) = 0.31

2. Primary Outcome: Physical Activity Hours Per Day Measured Using a Body-worn Accelerometer After 4 Months
Description: as for outcome 1
Time Frame: 4 months
Population: There were 2 participants lost to followup in both groups and 1 participant was missing accelerometer data in the control group. This results in a discrepancy with overall participant flow table which represents the number of participants with any available data.
Measure: Mean (Standard Deviation); unit: h/day
Arm/Group | Control | Treatment
Number analyzed (Participants) | 20 | 21
h/day | 1.5 (0.2) | 1.5 (0.2)
Statistical Analysis 1: Comparison: Control vs Treatment; Test type: Superiority; p = 0.78, Mixed Models Analysis — p-value is adjusted for multiple comparisons- P<0.025; controlled for baseline values as there was a significant difference between groups at baseline; Mean Difference (Final Values) = -0.02

3. Primary Outcome: Physical Activity Hours Per Day Measured Using a Body-worn Accelerometer After 6 Months
Description: as for outcome 1
Time Frame: 6 months
Population: 5 and 6 participants were lost to followup and additionally, accelerometer data were missing for 1 participant each in the control and treatment groups respectively. This results in a discrepancy with overall participant flow table which represents the number of participants with any available data.
Measure: Mean (Standard Deviation); unit: h/day
Arm/Group | Control | Treatment
Number analyzed (Participants) | 17 | 16
h/day | 1.5 (0.24) | 1.5 (0.24)
Statistical Analysis 1: Comparison: Control vs Treatment; Test type: Superiority; p = 0.56, Mixed Models Analysis — adjusted for multiple comparisons- P<0.025; controlled for baseline value due to a significant difference between groups at baseline; Mean Difference (Final Values) = 0.05

4. Primary Outcome: Sedentary Behavior Hours Per Day Measured Using a Body-worn Accelerometer at Baseline
Description: Total time spent sedentary will be measured using a body worn motion sensor (accelerometer) during waking hours over a period of one week. Measures for each day (hours) will be averaged to obtain a representative estimate of daily habitual behavior.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h/day
Arm/Group | Control | Treatment
Number analyzed (Participants) | 22 | 23
h/day | 10.6 (2.0) | 10.2 (2.0)
Statistical Analysis 1: Comparison: Control vs Treatment; Test type: Superiority; p = 0.4, Mixed Models Analysis; Mean Difference (Final Values) = -0.49

5. Primary Outcome: Sedentary Behavior Hours Per Day Measured Using a Body-worn Accelerometer After 4 Months
Description: as for outcome 4
Time Frame: 4 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h/day
Arm/Group | Control | Treatment
Number analyzed (Participants) | 20 | 21
h/day | 10.4 (1.9) | 9.6 (1.9)
Statistical Analysis 1: Comparison: Control vs Treatment; Test type: Superiority; p = 0.18, Mixed Models Analysis — p-value is adjusted for multiple comparisons and significance threshold was set at P<0.0167; Mean Difference (Final Values) = -0.80

6. Primary Outcome: Sedentary Behavior Hours Per Day Measured Using a Body-worn Accelerometer After 6 Months
Description: as for outcome 4
Time Frame: 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: h/day
Arm/Group | Control | Treatment
Number analyzed (Participants) | 17 | 16
h/day | 10.3 (1.8) | 10.2 (1.7)
Statistical Analysis 1: Comparison: Control vs Treatment; Test type: Superiority; p = 0.86, Mixed Models Analysis — p-value is adjusted for multiple comparisons and significance threshold was set at P<0.0167; Mean Difference (Final Values) = -0.11

7. Other Pre Specified Outcome: Percent Body Fat Measured Via Bioelectrical Impedance at Baseline
Description: This is an exploratory outcome. The amount of fat in the body will be computed as a percentage
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: % body fat
Arm/Group | Control | Treatment
Number analyzed (Participants) | 23 | 23
% body fat | 38.9 (5.8) | 41.1 (5.8)
Statistical Analysis 1: Comparison: Control vs Treatment; Test type: Superiority; p = 0.21, Mixed Models Analysis — p-value is adjusted for multiple comparisons and significance threshold was set at P<0.0167; Mean Difference (Final Values) = 2.2

8. Other Pre Specified Outcome: Percent Body Fat Measured Via Bioelectrical Impedance After 4 Months
Description: This is an exploratory outcome. The amount of fat in the body will be computed as a percentage
Time Frame: 4 months
Population: Missing data from 2 participants who were lost to follow-up in each group
Measure: Mean (Standard Deviation); unit: % body fat
Arm/Group | Control | Treatment
Number analyzed (Participants) | 21 | 21
% body fat | 38.2 (5.6) | 40.5 (5.6)
Statistical Analysis 1: Comparison: Control vs Treatment; Test type: Superiority; p = 0.19, Mixed Models Analysis — p-value is adjusted for multiple comparisons and significance threshold was set at P<0.0167; Mean Difference (Final Values) = 2.3

9. Other Pre Specified Outcome: Percent Body Fat Measured Via Bioelectrical Impedance After 6 Months
Description: This is an exploratory outcome. The amount of fat in the body will be computed as a percentage
Time Frame: 6 months
Population: 5 and 6 participants from the control and treatment group were lost to followup, respectively.
Measure: Mean (Standard Deviation); unit: % body fat
Arm/Group | Control | Treatment
Number analyzed (Participants) | 18 | 17
% body fat | 37.7 (5.2) | 40.5 (5.1)
Statistical Analysis 1: Comparison: Control vs Treatment; Test type: Superiority; p = 0.12, Mixed Models Analysis — p-value is adjusted for multiple comparisons and significance threshold was set at P<0.0167; Mean Difference (Final Values) = 2.8

10. Other Pre Specified Outcome: Attention and Executive Function Measured Using the NIH Tool Box Measured at Baseline
Description: This is an exploratory outcome - Average age-adjusted national percentile of NIH Toolbox Flanker Inhibitory Control and Attention Test score measured at Baseline. Each participant's raw score on the NIH Toolbox Flanker Inhibitory Control and Attention Test is standardized against a nationally representative sample to get the participant's national percentile. Percentiles are then adjusted for age and averaged across participants. Percentiles can range from 0 to 100, with a higher percentile indicating better performance.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: average age-adjusted percentile
Arm/Group | Control | Treatment
Number analyzed (Participants) | 23 | 23
average age-adjusted percentile | 36.2 (25.3) | 42.4 (25.3)
Statistical Analysis 1: Comparison: Control vs Treatment; Test type: Superiority; p = 0.41, Mixed Models Analysis — p-value is adjusted for multiple comparisons and significance threshold was set at P<0.0167; Mean Difference (Final Values) = 6.2

11. Other Pre Specified Outcome: Attention and Executive Function Measured Using the NIH Tool Box After 4 Months
Description: as for outcome 10
Time Frame: 4 months
Population: Two participants each were lost to follow-up in the control and treatment groups
Measure: Mean (Standard Deviation); unit: average age-adjusted percentile
Arm/Group | Control | Treatment
Number analyzed (Participants) | 21 | 21
average age-adjusted percentile | 46.0 (25.1) | 52.2 (25.5)
Statistical Analysis 1: Comparison: Control vs Treatment; Test type: Superiority; p = 0.43, Mixed Models Analysis — p-value is adjusted for multiple comparisons and significance threshold was set at P<0.0167; Mean Difference (Final Values) = 6.2

12. Other Pre Specified Outcome: Attention and Executive Function Measured Using the NIH Tool Box
Description: as for outcome 10
Time Frame: 6 months
Population: 5 and 6 participants from the control and treatment group were lost to followup, respectively.
Measure: Mean (Standard Deviation); unit: average age-adjusted score
Arm/Group | Control | Treatment
Number analyzed (Participants) | 18 | 17
average age-adjusted score | 50.3 (23.2) | 55.3 (23.8)
Statistical Analysis 1: Comparison: Control vs Treatment; Test type: Superiority; p = 0.53, Mixed Models Analysis — p-value is adjusted for multiple comparisons and significance threshold was set at P<0.0167; Mean Difference (Final Values) = 5.0

13. Other Pre Specified Outcome: Working Memory Measured Using the NIH Tool Box at Baseline
Description: This is an exploratory outcome - Average age-adjusted national percentile of NIH Toolbox Picture Sequence Memory Test score measured at Baseline. Each participant's raw score on the NIH Toolbox Picture Sequence Memory Test is standardized against a nationally representative sample to get the participant's national percentile. Percentiles are then adjusted for age and averaged accross participants. Percentiles can range from 0 to 100, with a higher percentile indicating better performance.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: average age-adjusted percentile
Arm/Group | Control | Treatment
Number analyzed (Participants) | 23 | 23
average age-adjusted percentile | 59.2 (28.8) | 59.0 (29.0)
Statistical Analysis 1: Comparison: Control vs Treatment; Test type: Superiority; p = 0.98, Mixed Models Analysis — p-value is adjusted for multiple comparisons and significance threshold was set at P<0.0167; Mean Difference (Final Values) = -0.17

14. Other Pre Specified Outcome: Working Memory Measured Using the NIH Tool Box After 4 Months
Description: This is an exploratory outcome - Average age-adjusted national percentile of NIH Toolbox Picture Sequence Memory Test score measured at Baseline. Each participant's raw score on the NIH Toolbox Picture Sequence Memory Test is standardized against a nationally representative sample to get the participant's national percentile. Percentiles are then adjusted for age and averaged across participants. Percentiles can range from 0 to 100, with a higher percentile indicating better performance.
Time Frame: 4 months
Population: Two participants each from the control and treatment group were lost to followup.
Measure: Mean (Standard Deviation); unit: average age-adjusted-percentile
Arm/Group | Control | Treatment
Number analyzed (Participants) | 21 | 21
average age-adjusted-percentile | 62.1 (28.2) | 61.7 (28.6)
Statistical Analysis 1: Comparison: Control vs Treatment; Test type: Superiority; p = 0.96, Mixed Models Analysis — p-value is adjusted for multiple comparisons and significance threshold was set at P<0.0167; Mean Difference (Final Values) = -0.47

15. Other Pre Specified Outcome: Working Memory Measured Using the NIH Tool Box After 6 Months
Description: as for outcome 14
Time Frame: 6 months
Population: 5 and 6 participants from the control and treatment group were lost to followup, respectively.
Measure: Mean (Standard Deviation); unit: average age-adjusted percentile
Arm/Group | Control | Treatment
Number analyzed (Participants) | 18 | 17
average age-adjusted percentile | 62.2 (26.1) | 63.3 (26.4)
Statistical Analysis 1: Comparison: Control vs Treatment; Test type: Superiority; p = 0.91, Mixed Models Analysis — p-value is adjusted for multiple comparisons and significance threshold was set at P<0.0167; Mean Difference (Final Values) = 1.1

16. Other Pre Specified Outcome: Relative Processing Speed Measured Using the NIH Tool Box at Baseline
Description: Average age-adjusted national percentile of NIH Toolbox Pattern Comparison Processing Speed Test score measured at Baseline. Each participant's raw score on the NIH Toolbox Pattern Comparison Processing Speed Test is standardized against a nationally representative sample to get the participant's national percentile. Percentiles are then adjusted for age and averaged across participants. Percentiles can range from 0 to 100, with a higher percentile indicating better performance.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Average age-adjusted percentile
Arm/Group | Control | Treatment
Number analyzed (Participants) | 23 | 23
Average age-adjusted percentile | 39.7 (38.2) | 52.7 (38.2)
Statistical Analysis 1: Comparison: Control vs Treatment; Test type: Superiority; p = 0.25, Mixed Models Analysis — p-value is adjusted for multiple comparisons and significance threshold was set at P<0.0167; Mean Difference (Final Values) = 13.1

17. Other Pre Specified Outcome: Relative Processing Speed Measured Using the NIH Tool Box Measured After 4 Months
Description: This is an exploratory outcome - Average age-adjusted national percentile of NIH Toolbox Pattern Comparison Processing Speed Test score measured at Baseline. Each participant's raw score on the NIH Toolbox Pattern Comparison Processing Speed Test is standardized against a nationally representative sample to get the participant's national percentile. Percentiles are then adjusted for age and averaged accross participants. Percentiles can range from 0 to 100, with a higher percentile indicating better performance.
Time Frame: 4 months
Population: Two participants each from the control and treatment group were lost to followup.
Measure: Mean (Standard Deviation); unit: Average age-adjusted percentile
Arm/Group | Control | Treatment
Number analyzed (Participants) | 21 | 21
Average age-adjusted percentile | 43.5 (37.1) | 52.0 (37.4)
Statistical Analysis 1: Comparison: Control vs Treatment; Test type: Superiority; p = 0.46, Mixed Models Analysis — p-value is adjusted for multiple comparisons and significance threshold was set at P<0.0167; Mean Difference (Final Values) = 8.5

18. Other Pre Specified Outcome: Relative Processing Speed Measured Using the NIH Tool Box Measured After 6 Months
Description: This is an exploratory outcome - Average age-adjusted national percentile of NIH Toolbox Pattern Comparison Processing Speed Test score measured at Baseline. Each participant's raw score on the NIH Toolbox Pattern Comparison Processing Speed Test is standardized against a nationally representative sample to get the participant's national percentile. Percentiles are then adjusted for age and averaged across participants. Percentiles can range from 0 to 100, with a higher percentile indicating better performance.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Average age-adjusted percentile
Arm/Group | Control | Treatment
Number analyzed (Participants) | 18 | 17
Average age-adjusted percentile | 49.0 (34.3) | 58.6 (34.3)
Statistical Analysis 1: Comparison: Control vs Treatment; Test type: Superiority; p = 0.41, Mixed Models Analysis — p-value is adjusted for multiple comparisons and significance threshold was set at P<0.0167; Mean Difference (Final Values) = 9.6

19. Other Pre Specified Outcome: Blood Glucose Measured Using a Cardiocheck Fingerstick Blood Sample Measured at Baseline
Description: This is an exploratory outcome.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control | Treatment
Number analyzed (Participants) | 23 | 23
mg/dL | 126.1 (30) | 112.3 (30)
Statistical Analysis 1: Comparison: Control vs Treatment; Test type: Superiority; p = 0.12, Mixed Models Analysis — p-value is adjusted for multiple comparisons and significance threshold was set at P<0.0167; Mean Difference (Final Values) = -13.8

20. Other Pre Specified Outcome: Blood Glucose Measured Using a Cardiocheck Fingerstick Blood Sample Measured After 4 Months
Description: This is an exploratory outcome.
Time Frame: 4 months
Population: Two participants each from the control and treatment group were lost to followup.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control | Treatment
Number analyzed (Participants) | 21 | 21
mg/dL | 127.7 (29.4) | 115.9 (29.4)
Statistical Analysis 1: Comparison: Control vs Treatment; Test type: Superiority; p = 0.20, Mixed Models Analysis — p-value is adjusted for multiple comparisons and significance threshold was set at P<0.0167; Mean Difference (Final Values) = -11.9

21. Other Pre Specified Outcome: Blood Glucose Measured Using a Cardiocheck Fingerstick Blood Sample Measured After 6 Months
Description: This is an exploratory outcome.
Time Frame: 6 months
Population: 5 and 6 participants from the control and treatment group were lost to followup, respectively.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control | Treatment
Number analyzed (Participants) | 18 | 17
mg/dL | 124.7 (27.2) | 110.7 (27.8)
Statistical Analysis 1: Comparison: Control vs Treatment; Test type: Superiority; p = 0.13, Mixed Models Analysis — p-value is adjusted for multiple comparisons and significance threshold was set at P<0.0167; Mean Difference (Final Values) = -14.0

22. Other Pre Specified Outcome: Total Cholesterol Measured Using a Cardiocheck Fingerstick Blood Sample Measured at Baseline
Description: This is an exploratory outcome.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control | Treatment
Number analyzed (Participants) | 23 | 23
mg/dL | 156.0 (41.3) | 156.8 (39.5)
Statistical Analysis 1: Comparison: Control vs Treatment; Test type: Superiority; p = 0.94, Mixed Models Analysis — p-value is adjusted for multiple comparisons and significance threshold was set at P<0.0167; Mean Difference (Final Values) = 0.83

23. Other Pre Specified Outcome: Total Cholesterol Measured Using a Cardiocheck Fingerstick Blood Sample Measured After 4 Months
Description: This is an exploratory outcome.
Time Frame: 4 months
Population: Two participants from the control and treatment group were lost to followup.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control | Treatment
Number analyzed (Participants) | 21 | 21
mg/dL | 161.0 (40.5) | 165.4 (38.6)
Statistical Analysis 1: Comparison: Control vs Treatment; Test type: Superiority; p = 0.72, Mixed Models Analysis — p-value is adjusted for multiple comparisons and significance threshold was set at P<0.0167; Mean Difference (Final Values) = 4.4

24. Other Pre Specified Outcome: Total Cholesterol Measured Using a Cardiocheck Fingerstick Blood Sample Were Measured After 6 Months
Description: This is an exploratory outcome.
Time Frame: 6 months
Population: 5 and 6 participants from the control and treatment group were lost to followup, respectively.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control | Treatment
Number analyzed (Participants) | 18 | 17
mg/dL | 152.9 (37.5) | 165.2 (36.4)
Statistical Analysis 1: Comparison: Control vs Treatment; Test type: Superiority; p = 0.33, Mixed Models Analysis — p-value is adjusted for multiple comparisons and significance threshold was set at P<0.0167; Mean Difference (Final Values) = 12.3

ADVERSE EVENTS:
Time Frame: Baseline, during face-to-face interactions, and after 4 and 16 weeks.
Arm/Group | Control | Treatment
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-03): https://cdn.clinicaltrials.gov/large-docs/12/NCT04827212/Prot_SAP_000.pdf